CLINICAL TRIAL: NCT06827860
Title: A Phase 2 Single-Arm Study of Subcutaneous Talquetamab in Elderly Patients With Multiple Myeloma in Early Relapse
Brief Title: Subcutaneous Talquetamab in Elderly Patients With Multiple Myeloma in Early Relapse
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Larysa Sanchez (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor-Investigator, Larysa Sanchez, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-00798; 64407564MMY2004 (Other: Janssen Research and Development)
Record Dates: First submitted 2025-02-03; First posted 2025-02-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Talquetemab; Elderly patients; Early relapse; Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — talquetamab; daratumumab

STUDY DESIGN:
Intervention Model Description: The study will utilize a Simon's two stage design with a total sample size of 23 patients. The study will start with a 28-day screening phase followed by a two-part treatment phase. In part 1, patients will receive talquetamab SC monotherapy starting with three step-up doses followed by the standard 800 μg/kg dose every other week. In part 2, participants will continue talquetamab and daratumumab until PD, unacceptable toxicity or other reasons for discontinuing treatment, withdrawal from study. Patients in part 1 and part 2 who achieve VGPR or better after receiving at least 4 cycles of talquetamab in the respective part can be transitioned to every 4 week dosing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Talquetamab SC monotherapy (Experimental): In part 1, patients will receive talquetamab SC monotherapy starting with three step-up doses followed by the standard 800 μg/kg dose every other week. Cycles will be 28 days long. Response will be assessed monthly according to IMWG criteria, and patients who have PD after completing at least 1 cycle of talquetamab or who fail to attain ≥ PR after completion of cycle 3 will proceed to part 2 only if not previously refractory to an anti-CD38 monoclonal antibody. Patients refractory to an anti-CD38 mAb will not be allowed in Part 2. patients who are refractory to an anti-CD38 mAb and PD at any point will be taken off study and not proceed to Part 2. patients who are refractory to an anti-CD38 mAb and achieve a response <PR after 3 cycles (stable disease or minimal response) will continue on talquetamab monotherapy until PD or be taken off study per investigator discretion if it is deemed that subject will not continue to derive clinical benefit from talquetamab monotherapy.
  Interventions: Drug: Talquetamab
- Talqeutemab SC + Daratumumab SC (Experimental): For participants who proceed to part 2, talquetamab will be continued at 800 μg/kg every other week but daratumumab will be initiated at the standard dose (weekly for 2 cycles, every other week for 4 cycles, monthly thereafter). In part 2, participants will continue talquetamab and daratumumab until PD, unacceptable toxicity or other reasons for discontinuing treatment, withdrawal from study. Patients in part 1 and part 2 who achieve VGPR or better after receiving at least 4 cycles of talquetamab in the respective part can be transitioned to every 4 week dosing.
  Interventions: Drug: Talquetamab; Drug: Daratumumab

INTERVENTIONS:
Drug: Talquetamab — SC monotherapy starting with three step-up doses followed by the standard 800 μg/kg dose every other week. Cycles will be 28 days long.
  Other Names: JNJ-64407564
Drug: Daratumumab — SC at the standard dose (weekly for 2 cycles, every other week for 4 cycles, monthly thereafter)
  Arms: Talqeutemab SC + Daratumumab SC

SUMMARY:
Induction therapy approaches in recent years have evolved, now utilizing triple or quadruple drug regimens in the majority of patients. By combining anti-CD38 antibodies, proteasome inhibitors (PIs), immunomodulatory drugs (IMiDs), and steroids, patients achieve longer remissions with their first- and second-line therapies but also become refractory to most or all three major drug classes earlier. For patients who are refractory to at least 3 of the commonly administered PIs and IMiDs, occurring after 2 lines of therapy in many, the median overall survival is only 5 months. Elderly, frail patients are not often candidates at this point for aggressive therapies like stem cell transplantation and CAR T-cell therapy thus necessitating effective yet tolerable treatments for elderly patients in early relapse (1-3 prior therapy). Talquetamab is a GPRC5DxCD3 bispecific antibody that redirects patients' T cells to myeloma cells which express GPRC5D. In the phase 1 MonumenTAL-1, heavily pretreated patients with a median of 6 prior lines of therapy attained a 70% response rate with 405 μg/kg of subcutaneous (SC) talquetamab. Importantly, subcutaneous talquetamab was found to be tolerable for the treated population, which included 28% of patients aged ≥70, with only three patients experiencing dose-limiting toxicities in the form of grade 3 rashes which responded to steroids. The anti-CD38 antibody daratumumab eliminates CD38-positive T and B regulatory cells, potentiates the activity of bispecific antibodies like talquetamab, and may improve its efficacy when used in combination. The aim of this study will be to assess the efficacy and safety of treating elderly patients with relapsed/refractory multiple myeloma with at least ≥2 prior lines of therapy with subcutaneous talquetamab. Patients who have progressive disease on talquetamab or who fail to respond after 3 cycles will have subcutaneous daratumumab added to their regimen.

ELIGIBILITY:
Inclusion Criteria:

* Documented multiple myeloma as defined by the criteria below:

  * Multiple myeloma diagnosis according to the IMWG diagnostic criteria
  * Measurable disease at screening as assessed by central laboratory, defined by at least 1 of the following:
* Serum M-protein level ≥0.5 g/dL (central laboratory)
* Urine M-protein level ≥200 mg/24 hours (central laboratory)
* Light chain multiple myeloma without measurable M-protein in the serum or the urine: serum immunoglobulin free light chain ≥10 mg/dL or >100 mg/L (central laboratory) provided the serum free light chain ratio is abnormal (0.22 to 1.52 [central laboratory])

NOTE: Local laboratory results of blood and urine M-protein measurements may be used to determine initial eligibility. Central laboratory results should still be obtained prior to the start of administration of study treatment in order to establish baseline values and confirm the results from the local laboratory.

• Relapsed or refractory disease as defined below:

* Relapsed disease is defined as an initial response to prior treatment, followed by confirmed progressive disease by IMWG criteria >60 days after cessation of treatment.
* Refractory disease is defined as <25% reduction in M-protein or confirmed progressive disease by IMWG criteria during previous treatment or ≤60 days after cessation of treatment. Received at least 1 prior line(s) of antimyeloma therapy including a minimum of 2 consecutive cycles

NOTE: Participant must have undergone ≥1 complete cycle of treatment for each regimen, unless progressive disease was the best response to the regimen.

NOTE: A single line of therapy may consist of 1 or more agents and may include induction, hematopoietic stem cell transplantation, and maintenance therapy. Radiotherapy, bisphosphonate, or a single short course of corticosteroids (no more than the equivalent of dexamethasone 40 mg/day for 4 days) would not be considered prior lines of therapy.

* Subject must have received at least ≥2 prior line(s) of systemic antimyeloma therapy of treating physician's discretion, including a PI and an IMID
* Subjects who are anti-CD38 monoclonal antibody-naïve, exposed, or refractory will be allowed in Part 1; Only subjects who are anti-CD38 antibody-naïve or exposed will be allowed in Part 2, whereas subjects refractory to anti-CD38 monoclonal antibody will not be allowed in Part 2
* Have clinical laboratory values meeting the following criteria during the Screening Phase: Hematology Hemoglobin: ≥7 g/dL (≥4.96 mmol/L; without transfusion support or erythropoietin use within 7 days before the laboratory test) Platelets: ≥50×109/L (without transfusion support or thrombopoietin receptor agonist within 7 days before the laboratory test) Absolute neutrophil count: ≥1.0×109/L (prior growth factor support is permitted but must be without support for 7 days for G-CSF or GM-CSF and for 14 days for pegylated GCSF before the laboratory test) Chemistry AST and ALT: ≤2.5×ULN eGFR: ≥30 mL/min based on Modified Diet in Renal Disease Formula calculation Total bilirubin: ≤2.0×ULN; except in participants with congenital bilirubinemia, such as Gilbert syndrome (in which case direct bilirubin ≤1.5×ULN is required) Serum calcium corrected for albumin: ≤14 mg/dL (≤3.5 mmol/L) or free ionized calcium ≤6.5 mg/dL (≤1.6 mmol/L;)
* Human immunodeficiency virus-positive participants are eligible if they meet all of the following:

  * No detectable viral load (ie, <50 copies/mL) at screening
  * CD4+ count >300 cells/mm3 at screening
  * No acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within 6 months of screening
  * Receiving HAART. Any changes in HAART due to resistance/progression should occur at least 3 months prior to screening. A change in HAART due to toxicity is allowed up to 4 weeks prior to screening.

Note: HAART that could interfere with study treatment is excluded (consult the sponsor for a review of medications prior to enrollment) • A male participant must agree to wear a condom (with spermicidal foam/gel/film/cream/suppository) when engaging in any activity that allows for passage of ejaculate to another person during the study and for a minimum of 100 days after receiving the last dose of study treatment.

NOTE: If the male participant is vasectomized, he still must wear a condom (with foam/gel/film/cream/suppository), but his female partner is not required to use contraception.

* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 100 days after receiving the last dose of study treatment.
* Must be willing and able to adhere to the prohibitions and restrictions specified in this protocol (Section 2, including to not donate blood or blood components during the study and for 100 days after the last dose of study drug)
* Sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study, and is willing to and able to participate in the study. Consent is to be obtained prior to the initiation of any study-related tests or procedures that are not part of standard-of-care for the subject's disease.

Exclusion Criteria:

Any potential subject who meets any of the following criteria will be excluded from participating in the study:

* Contraindications or life-threatening allergies, hypersensitivity, or intolerance to any study drug or its excipients (refer to the talquetamab and daratumumab Investigator's Brochure and appropriate prescribing information).
* Prior treatment with T-cell-engaging antibodies
* Prior antitumor therapy as follows, prior to the first dose of study drug:

  o Any prior GPRC5D-directed therapy
  * Gene-modified adoptive cell therapy (eg, chimeric antigen receptor modified T cells, NK cells) within 3 months
  * Targeted therapy, epigenetic therapy, or treatment with an investigational drug or an invasive investigational medical device within 21 days or at least 5 half-lives, whichever is less.
  * Investigational vaccine other than SARS CoV-2 vaccine approved/ in use under emergency approval within 4 weeks o Live, attenuated vaccine within 4 weeks
  * Monoclonal antibody treatment for multiple myeloma within 21 days.
  * Cytotoxic therapy within 21 days.
  * Proteasome inhibitor therapy within 14 days. o Immunomodulatory agent therapy within 14 days. o Radiotherapy within 14 days or focal radiation within 7 days
* Toxicities from previous anticancer therapies should have resolved to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy.
* Received a maximum cumulative dose of corticosteroids equivalent to ≥140 mg of prednisone within the 14-day period before the first dose of study drug.
* Stem cell transplantation:

  * Previous allogenic stem cell transplant
  * Received an autologous stem cell transplant ≤12 weeks before the first dose of study drug
* Known active CNS involvement or exhibits clinical signs of meningeal involvement of multiple myeloma. If either is suspected, negative whole brain MRI and lumbar cytology are required.
* Plasma cell leukemia (>20% circulating plasma cells and/or >2.0 x 109/L plasma cells by standard differential), Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein [M-protein], and skin changes), or primary amyloid light chain amyloidosis.
* Myelodysplastic syndrome or active malignancies (ie, progressing or requiring treatment change in the last 24 months) other than relapsed/refractory multiple myeloma. The only allowed exceptions are:

  o Non-muscle invasive bladder cancer treated within the last 24 months that is considered completely cured

  o Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured
  * Noninvasive cervical cancer treated within the last 24 months that is considered completely cured
  * Localized prostate cancer (N0M0):

    - With a Gleason score of ≤6, treated within the last 24 months, or untreated and under surveillance
    * With a Gleason score of 3+4 that has been treated >6 months prior to full study screening and considered to have a very low risk of recurrence, or
    * History of localized prostate cancer and receiving androgen deprivation therapy and considered to have a very low risk of recurrence
  * Breast cancer: adequately treated lobular carcinoma in situ or ductal carcinoma in situ, or history of localized breast cancer and receiving antihormonal agents and considered to have a very low risk of recurrence
  * Other malignancy that is considered cured with minimal risk of recurrence.
* Stroke or seizure within 6 months prior to signing ICF.
* Any of the following:

  * Active Hepatitis B infection (ie, HBsAg or HBV-DNA positive). In the event the infection status is unclear, quantitative viral levels are necessary to determine the infection status see Section Hepatitis B Virus Testing 8.7.1.18.7.1 for further required assessments.
  * Active hepatitis C infection as measured by positive HCV-RNA testing. Participants with a history of HCV antibody positivity must undergo HCV-RNA testing. If a participant with history of chronic hepatitis C infection (defined as both HCV antibody and HCV-RNA positive) completed antiviral therapy and has undetectable HCV-RNA for at least 12 weeks following the completion of therapy, the participant is eligible for the study.
* Any concurrent medical or psychiatric condition or disease that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study, such as:

  * Uncontrolled diabetes o Acute diffuse infiltrative pulmonary disease
  * Evidence of active systemic viral, fungal, or bacterial infection, requiring systemic antimicrobial therapy within 7 days of start of study treatment
  * Active autoimmune disease requiring systemic immunosuppressive therapy within 6 months before start of study treatment.

EXCEPTION: Participants with vitiligo, controlled type I diabetes, and prior autoimmune thyroiditis that is currently euthyroid based on clinical symptoms and laboratory testing are eligible regardless of when these conditions were diagnosed.

* Disabling psychiatric conditions (e.g., alcohol or drug abuse), severe dementia, or altered mental status
* Any other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site, to understand informed consent or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* History of non-compliance with recommended medical treatments • Plans to father a child while enrolled in this study or within 100 days after the last dose of study drug.

  • Presence of the following cardiac conditions:
* New York Heart Association stage III or IV congestive heart failure
* Myocardial infarction or coronary artery bypass graft ≤6 months prior to randomization
* Uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities
* History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration o History of severe non-ischemic cardiomyopathy • Major surgery within 2 weeks prior to the start of administration of study treatment, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to be treated in the study or within 2 weeks after administration of the last dose of study treatment.
* NOTE: Participants with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery. If there is a question whether a procedure is considered a major surgery, the investigator must consult with the appropriate sponsor representative and resolve any issues before enrolling a participant in the study • Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal of DLCO <50%).

Note: FEV1 testing is required for participants suspected of having COPD and participants must be excluded if FEV1 <50% of predicted normal.

• Known moderate of persistent asthma within the past 2 years or currently has uncontrolled asthma of any classification.

Note: Participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study.

NOTE: Investigators should ensure that all study inclusion/exclusion criteria have been met at screening and prior to the first dose of study drug. If a subject's clinical status changes (including any available laboratory results or receipt of additional medical records) after screening but before the first dose of study drug is given such that he or she no longer meets all eligibility criteria, supportive treatment may be administered according to local standards of care, if necessary, so that eligibility criteria may be met and laboratory test(s) may be repeated once, to determine if the subject qualifies for the study. If inclusion/exclusion criteria are not met after further evaluation, the subject should be excluded from participation in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Completion of part 1 of the study after completion of 3 cycles (each cycle is 28 days each) or until PD, whichever occurs first.
  ORR defined as the proportion of patients who achieve ≥PR according to IMWG criteria in the intention-to-treat population in Part 1

SECONDARY OUTCOMES:
Time to progression (TTP) for talquetamab monotherapy | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  Time to progression (TTP) defined as the duration from the first date of study treatment to the date of first documented evidence of PD or death in Part 1, whichever comes first
Progression-free survival (PFS) for talquetamab monotherapy | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  PFS defined as the duration from the first date of study treatment to the date of first documented evidence of PD or death in Part 1, whichever comes first
Overall survival (OS) for talquetamab monotherapy | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  OS defined as the duration from the first date of study treatment to the date of the subject's death
Duration of response (DOR) for talquetamab monotherapy | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  DOR defined as the duration from the date of initial attainment of ≥PR to first documented evidence of progressive disease (PD) in Part 1
ORR2 with addition of daratumumab | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  ORR2 defineORR2d as the proportion of patients who achieve ≥PR according to IMWG criteria in Part 2
DOR2 with addition of daratumumab | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  DOR2 defined as the duration from the date of initial attainment of ≥PR to first documented evidence of progressive disease (PD) in Part 2.
PFS2 with addition of daratumumab | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  PFS2 defined as the duration from first treatment with daratumumab in Part 2 to PD or death
ORR2 for talquetamab monotherapy and in combination with daratumumab | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  ORR2 defined as the proportion of patients who achieve ≥PR according to IMWG criteria in Part 2
DOR2 for talquetamab monotherapy and in combination with daratumumab | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  DOR2 defined as the duration from the date of initial attainment of ≥PR to first documented evidence of progressive disease (PD) in Part 2.
PFS2 for talquetamab monotherapy and in combination with daratumumab | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  PFS2 defined as the duration from first treatment with daratumumab in Part 2 to PD or death
Number of participants with response evaluation criteria of talquetamab monotherapy and in combination with daratumumab | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  Number of participants with response evaluation criteria of talquetamab monotherapy and in combination with daratumumab using stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), minimal residual disease (MRD) negativity,
Clinical benefit rate (CBR) for talquetamab monotherapy and in combination with daratumumab | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  Clinical benefit rate (CBR)
Time to ORR for talquetamab monotherapy and in combination with daratumumab | Evaluated continuously until end of study (due to disease progression or death from any cause, whichever comes first), assessed up to 36 months
  Time to ORR (≥PR), ≥VGPR, ≥CR, and sCR and MRD negativity, defined as the duration from the date of initial therapy to the date of attainment of a response category and was subsequently confirmed by a repeated measurement as required by the IMWG criteria
Myeloma Patient Outcomes Scale (MyPOS) | Baseline, C4D1 (cycle 4 day 1), and C13D1 (cycle 13 day 1), each cycle is 28 days each
  To assess quality of life (QOL) on talquetamab using the Myeloma Patient Outcomes Scale (MyPOS).
  Full scale from 0-100, with higher scores representing worse QOL

CONTACTS AND LOCATIONS:
Overall Officials: Larysa Sanchez, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link tbd).